CLINICAL TRIAL: NCT02949947
Title: Efficacy of Ferric Carboxymaltose in Gastrointestinal Stromal Tumor (GIST) Patients With Iron Deficiency Anemia (IDA) Receiving Systemic Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated per PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0588; NCI-2016-01925 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Malignant Neoplasms of Mesothelial and Soft Tissue; Gastrointestinal Stromal Tumor With Neurogenic Differentiation
Keywords: Malignant Neoplasms of Mesothelial and Soft Tissue; Gastrointestinal Stromal Tumor; GIST; Iron-deficiency anemia; Ferric Carboxymaltose; Injectafer; Iron supplement; Health Questionnaire; Survey
MeSH Terms: conditions — Plexosarcoma; Gastrointestinal Stromal Tumors; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Iron-Dextran Complex; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - Ferric Carboxymaltose (Experimental): Participants receive a Ferric Carboxymaltose injection by vein. Dose repeated 1 week later.
  Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
  Interventions: Drug: Ferric Carboxymaltose; Behavioral: Questionnaire
- Group B - Iron Supplement (Active Comparator): Participants take iron supplements by mouth every day for up to 3 months.
  Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
  Interventions: Dietary Supplement: Iron Supplements; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Ferric Carboxymaltose — 15 mg/kg by vein (up to 750 mg) over 15 min infusion. Dose repeated 1 week later.
  Other Names: Injectafer
  Arms: Group A - Ferric Carboxymaltose
Dietary Supplement: Iron Supplements — Participants take iron supplements by mouth every day for up to 3 months.
  Arms: Group B - Iron Supplement
Behavioral: Questionnaire — Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to compare Injectafer® (ferric carboxymaltose) with an iron supplement to learn which may be more effective in improving red blood cell counts in patients who have iron-deficiency anemia (a low red blood cell count) because of a gastrointestinal stromal tumor (GIST) and/or systemic therapy.

The safety of ferric carboxymaltose will also be studied.

This is an investigational study. Ferric carboxymaltose is FDA approved and commercially available to treat iron deficiency anemia; however, it is considered investigational to use in patients who have cancer-related or systemic therapy-related anemia.

Up to 50 participants will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one group is better, the same, or worse than the other.

* If you are in Group A, you will receive ferric carboxymaltose injection by vein over about 15 minutes. You will receive 2 injections about 7 days apart (for example, on Days 0 [the day you are assigned to a study group] and 7).
* If you are in Group B, you will take iron supplements by mouth every day. This is considered standard of care for iron deficiency anemia and the study staff will discuss with you which iron supplements you will take and their risks.

You and the study staff will know to which group you are assigned.

Length of Study:

You may receive up to 2 injections of ferric carboxymaltose (if you are in Group A) or up to 3 months of oral iron supplements (if you are in Group B). You will no longer be able to take the study drug if intolerable side effects occur or if you are unable to follow study directions.

Your participation on the study will be over after you have completed the Week 24 visit.

Study Visits:

Baseline (within 1 week after you have been assigned to a study group):

* You will have a physical exam.
* You will complete a questionnaire about your health. It should take about 5 minutes to complete.
* Blood (about 1 tablespoon) will be drawn for routine tests and to test the level of iron in your blood.

One (1) time every week during Months 1-3, blood (about 1 tablespoon) will be drawn for routine tests.

At about Weeks 4, 8, 12, and 24 (the end-of-study visit):

* You will have a physical exam (Weeks 12 and 24 only).
* You will complete the same questionnaire you did at baseline.
* Blood (about 1 tablespoon) will be drawn for routine tests and to test the level of iron in your blood.

During Weeks 16 and 20, blood (less than 1 tablespoon) will be drawn to test the level of iron in your blood.

If you leave the study before Week 24, you will have the Week 24 study visits as soon as possible after you leave the study.

ELIGIBILITY:
Inclusion Criteria:

1. GIST patients with IDA planned to start or are receiving systemic therapy with TKIs.
2. Evidence of iron deficiency anemia including, Hgb < 11 g/dL, but > 8 g/dL; and transferrin saturation (TSAT) < 20%.
3. No H/O allergic reaction to iron therapy.
4. No clinical signs active of bleeding.
5. Adequate hematologic (ANC > 1500/mm^3, platelet count > 100,000/mm^3), renal (serum creatinine < 1.5mg/dL), and hepatic (serum bilirubin count < 1.5 x normal and serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) < 3 x normal) functions.
6. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
7. Signed informed consent to the study.
8. Male and Females of child bearing potential must use acceptable methods of birth control which include oral contraceptives, spermicide with either a condom, diaphragm or cervical cap, use of an intrauterine device (IUD) or abstinence.
9. Patients are required to read and understand English to comply with protocol requirements.
10. Age >=18 years old.
11. Life expectancy of at least 6 months.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with any co-morbid condition which renders patients at high risk of treatment complication.
3. Patient has uncontrolled angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%), uncontrolled cardiac arrhythmia or hypertension, or acute myocardial infarction within 3 months.
4. Patient has an active seizure disorder. (Patients with a previous history of seizure disorders will be eligible for the study, if they have had no evidence of seizure activity, and they have been free of antiseizure medication for the previous 5 years).
5. Psychological, social, familial, or geographical reasons that would prevent scheduled visits and follow-up.
6. Prior surgery or radiotherapy (RT) within 2 weeks of study entry.
7. Known hypersensitivity reaction to any component of ferric carboxymaltose.
8. Any anemia treatment within 4 weeks before inclusion (oral iron, IV iron, or erythropoiesis-stimulating agents), or transfusion of PRBCs in 2 weeks.
9. Hemochromatosis or other iron storage disorders.
10. Known positive hepatitis with evidence of active disease.
11. Patients with overt bleeding.
12. Ferritin >/= 800 ng/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 12/2017 to 1/2019
Pre-assignment Details: A total of 3 participants were enrolled in the study; however only 1 started on the trial since 1 participant non-compliance and 1 participant insurance changed. Due to low accrual the study terminated early.
Groups:
- Group A - Ferric Carboxymaltose: Participants receive a Ferric Carboxymaltose injection by vein. Dose repeated 1 week later.
  Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
  Ferric Carboxymaltose: 15 mg/kg by vein (up to 750 mg) over 15 min infusion. Dose repeated 1 week later.
  Questionnaire: Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
- Group B - Iron Supplement: Participants take iron supplements by mouth every day for up to 3 months.
  Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
  Iron Supplements: Participants take iron supplements by mouth every day for up to 3 months.
  Questionnaire: Health questionnaire completed at Baseline and at Weeks 4, 8, 12, and 24.
Period: Overall Study
Arm/Group | Group A - Ferric Carboxymaltose | Group B - Iron Supplement
Started | 1 | 2
Completed | 0 | 1
Not Completed | 1 | 1
Not completed — Non Compliance | 0 | 1
Not completed — Insurance change | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Ferric Carboxymaltose | Group B - Iron Supplement | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate in Hemoglobin (HGB)
Description: The primary endpoint is response (CR rate) in HGB within 3 months. Participant considered as to have a complete response (CR) if his/her HGB level increases > 2 g/dL from baseline during 3 months following initiation of the study drug, and/or transfusion-dependent patient is transfusion free.
Time Frame: 3 months
Population: Due to early termination of the protocol and low accrual not enough data collected to analyze the Complete Response Rate in Hemoglobin.
Arm/Group | Group A - Ferric Carboxymaltose | Group B - Iron Supplement
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 3 months
Arm/Group | Group A - Ferric Carboxymaltose | Group B - Iron Supplement
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Ferric Carboxymaltose (N=1) | Group B - Iron Supplement (N=2)
Constipation (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT02949947/Prot_SAP_000.pdf